CLINICAL TRIAL: NCT04403516
Title: Dextenza in Pterygium Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Michelle Rhee MD (Other)
Collaborators: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Michelle Rhee MD, Principal Investigator, New York Eye Specialists
Organization: New York Eye Specialists (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dextenza in Pterygium Surgery
Record Dates: First submitted 2020-05-12; First posted 2020-05-27 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Pterygium
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Intervention Model Description: In patients who undergo pterygium surgery, eyes will be consecutively assigned to receive either DEXTENZA (15 eyes) into both the upper and lower puncta at the time of surgery, followed by at postoperative month 1 visit institution of topical prednisolone acetate 1% bid x 2 weeks then qd x 2 weeks then discontinued or receive topical prednisolone acetate 1% (15 eyes) q2 hours x 2 weeks then qid for 2 weeks then bid for 2 weeks then qd for 2 weeks then discontinued.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- DEXTENZA Group (Experimental): Patients with Pterygium DEXTENZA Group
  Interventions: Drug: Dexamethasone Intracanalicular Insert, 0.4mg
- Topical Prednisolone Acetate 1% Group (Experimental): Patients with Pterygium Topical Prednisolone Acetate 1% Group
  Interventions: Drug: Prednisolone Acetate 1%

INTERVENTIONS:
Drug: Dexamethasone Intracanalicular Insert, 0.4mg — To determine post-surgical resolution of pain and inflammation outcomes with DEXTENZA compared to topical steroid treatment in patients who undergo pterygium surgery.
  Arms: DEXTENZA Group
Drug: Prednisolone Acetate 1% — To reduce post-surgical pain and inflammation in patients who undergo pterygium surgery.
  Arms: Topical Prednisolone Acetate 1% Group

SUMMARY:
DEXTENZA for the treatment of post-surgical pain and inflammation compared to standard of care topical prednisolone acetate 1% in patients who undergo pterygium surgery (excision of pterygium with conjunctival autograft)

DETAILED DESCRIPTION:
In patients who undergo pterygium surgery, eyes will be consecutively assigned to receive either DEXTENZA or topical prednisolone acetate 1%.15 eyes will receive a Dextenza insertion into both the upper and lower puncta at the time of surgery, followed by at postoperative month 1 visit institution of topical prednisolone acetate 1% bid x 2 weeks then qd x 2 weeks then discontinued. 15 eyes will receive starting on postoperative day 1 topical prednisolone acetate 1% q2 hours x 2 weeks then qid for 2 weeks then bid for 2 weeks then qd for 2 weeks then discontinued.

ELIGIBILITY:
Inclusion Criteria:

A patient's study eye must meet the following criteria to be eligible for inclusion in the study:

• Age of at least 18 years with primary pterygia

Exclusion Criteria:

A patient who meets any of the following criteria will be excluded from the study:

* Glaucoma
* Ocular hypertension
* Prior conjunctival surgery
* Other uncontrolled ocular disease
* Ocular surgery in either eye within 3 months
* Use of eye drops other than postoperative medications and artificial tears

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-05 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction-comfort and convenience | Assessed on Post-Op Day 1
  Assessed by patient reported questionnaire
Patient satisfaction-comfort and convenience | Assessed on Week 1
  Assessed by patient reported questionnaire
Patient satisfaction-comfort and convenience | Assessed on Month 1
  Assessed by patient reported questionnaire
Patient satisfaction-comfort and convenience | Assessed on Month 3
  Assessed by patient reported questionnaire
Patient satisfaction-comfort and convenience | Assessed on Month 6
  Assessed by patient reported questionnaire

SECONDARY OUTCOMES:
To compare the degree of conjunctival hyperemia | Assessed on Week 1
  Assessed by clinical external photography
To compare the degree of conjunctival hyperemia | Assessed on Month 1
  Assessed by clinical external photography
To compare the degree of conjunctival hyperemia | Assessed on Month 2
  Assessed by clinical external photography
To compare the degree of conjunctival hyperemia | Assessed on Month 3
  Assessed by clinical external photography
To compare the degree of conjunctival hyperemia | Assessed on Month 6
  Assessed by clinical external photography
Mean number of days for corneal re-epithelialization | Assessed on Post-Op Day 1
  As evaluated by slit lamp examination
Mean number of days for corneal re-epithelialization | Assessed on Week 1
  As evaluated by slit lamp examination
Mean number of days for corneal re-epithelialization | Assessed on Month 1
  As evaluated by slit lamp examination
Recurrence of pterygium | Assessed at Month 1
  As measured by yes or no on recurrence; external eye examination
Recurrence of pterygium | Assessed at Month 2
  As measured by yes or no on recurrence; external eye examination
Recurrence of pterygium | Assessed at Month 3
  As measured by yes or no on recurrence; external eye examination
Recurrence of pterygium | Assessed at Month 6
  As measured by yes or no on recurrence; external eye examination

CONTACTS AND LOCATIONS:
Overall Officials: Michelle K Rhee, MD, Principal Investigator — New York Eye Specialists
Locations (1):
- New York Eye Specialists, New York, New York, United States

REFERENCES:
- [Derived] Rhee MK, Zakher M, Najac M, Arias H, Jo J, Gorham R, Moadel K. Comparing Intracanalicular and Topical Steroid Use in Patients Undergoing Pterygium Surgery. Eye Contact Lens. 2024 Apr 1;50(4):183-188. doi: 10.1097/ICL.0000000000001075. Epub 2024 Feb 1. PMID 38305478